CLINICAL TRIAL: NCT03879629
Title: TrAstuzumab Cardiomyopathy Therapeutic Intervention With Carvedilol (TACTIC) Trial
Brief Title: Treating Breast Cancer Patients Undergoing Trastuzumab Treatment With Carvedilol to Reduce Incidence of Heart Failure
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Miami Heart Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TACTIC; R01CA233610 (NIH); NCI-2019-08427 (Other Grant/Funding Number: NCI); MC1932 (Other: Mayo Clinic); 18-006090 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-03-08; First posted 2019-03-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pre-Emptive Strategy (Experimental): Carvedilol titrated to maximally tolerated doses (3.125 mg to 25 mg twice a day) initiated one week before start of therapy and continued until end of therapy
  Interventions: Drug: Carvedilol
- Reactive Strategy (Experimental): Carvedilol titrated to maximally tolerated doses (3.125 mg to 25 mg twice a day) initiated after documentation of subclinical cardiotoxicity, defined by an abnormal global longitudinal strain (GLS) or high-sensitive cardiac troponin (hsTnI) elevation and continued until end of therapy
  Interventions: Drug: Carvedilol
- Standard of Care (Active Comparator): Carvedilol titrated to maximally tolerated doses (3.125 mg to 25 mg twice a day) initiated after documentation of a drop in LVEF by >10% to a value less than 53% and continued until end of therapy
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — oral Carvedilol maximally tolerated doses 3.125 mg to 25 mg twice a day
  Other Names: Coreg

SUMMARY:
Breast cancer patients undergoing trastuzumab-based HER2-directed therapy are at risk of heart function decline or heart failure symptoms, but it is unknown if, when, and for how long cardiovascular protective strategies, e.g. with a beta-blocker, could help. This study randomly assigns those taking curative-intent trastuzumab-based HER2-directed therapy to the beta-blocker carvedilol-either when significant heart function decline or subtle early signs of heart injury (either by elevation of a cardiac blood biomarker, i.e. cardiac troponin, or by an abnormal heart ultrasound marker, i.e. global longitudinal strain) are noted, or preventatively before beginning trastuzumab-based HER2-directed therapy. This study will further randomly assign those patients on carvedilol to either discontinuation at the end of trastuzumab-based HER2-directed therapy or continuation for another year, providing much needed clinical trial data on what the best strategy ("tactic") for those at risk of cardiotoxicity with trastuzumab-based HER2-directed therapy is.

DETAILED DESCRIPTION:
The objective of the current application is to evaluate different strategies of cardiovascular therapy with carvedilol, aiming to reduce the incidence of LVEF decline and HF in patients undergoing curative intent trastuzumab-based HER2-directed therapy for breast cancer. It will compare: a) a pre-emptive preventive approach, i.e. cardiovascular therapy with the beta-blocker carvedilol started before trastuzumab-based HER2-directed therapy and b) a reactive preventive approach, i.e. cardiovascular therapy started in response to early subclinical signs of cardiac dysfunction/injury (either cardiac troponin elevation or abnormal global longitudinal strain), with the current standard approach of initiation cardiovascular therapy once cardiotoxicity has occurred, addressing the question if and at which point in time carvedilol therapy would be efficacious. It will furthermore compare outcome measures between a limited carvedilol therapy duration, confined to the time of the active trastuzumab-based HER2-directed treatment and cardiac function recovery versus an extended carvedilol therapy duration continuing one year after completion of trastuzumab-based HER2-directed therapy, addressing how long carvedilol needs to be given in this unique patient population. The above will be combined with pharmacogenomic measures to identify those at highest risk of irreversible LVEF decline and lack of response to therapy. The investigator's central hypothesis is that a pre-emptive or a reactive preventive approach will reduce the incidence of cardiotoxicity in breast cancer patients undergoing treatment with trastuzumab, and that extension of carvedilol therapy beyond the active trastuzumab-based HER2-directed therapy treatment will prove superior for preservation of cardiac function.

Three specific aims will be pursued:

Aim 1: to compare the incidence of a) HF or asymptomatic decline in LVEF by >10% in patients whose LVEF is ≥50% or LVEF drop ≥5% in those with a decrease to <50%. (primary aim #1), and b) reversible LVEF decline to within 5% of baseline (secondary aim #1) with a pre-emptive and reactive preventive approach with carvedilol versus a "wait-and-see strategy" of carvedilol initiation in response to HF or LVEF declines in breast cancer patients over the course of trastuzumab therapy. It is to address the question if and when to start cardioprotective efforts for patients undergoing trastuzumab therapy.

Aim 2: To compare the delta change in LVEF from completion to one year after completion of trastuzumab therapy between cardioprotective approach with carvedilol confined the duration of trastuzumab therapy or extended for one year thereafter. This aim is to address the question of duration of cardioprotective efforts for patients undergoing trastuzumab therapy.

Aim 3: To identify genetic variants that predict trastuzumab cardiotoxicity in general as well as lack of response (primary prevention of drop in LVEF or secondary improvement of LVEF) to carvedilol.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age,
* new or locally recurrent diagnosis of HER2+ breast cancer that will be treated with curative intent
* planned HER2-directed (any therapy targeting HER2 signaling including Trastuzumab +/- pertuzumab or trastuzumab-emtansine (T-DM1) Nerantinib and lapatinib will not be considered. "HER2-directed therapy" or "anti-HER-2".

Exclusion Criteria:

* history of HF of any class and type, or diagnosis of cardiomyopathy in the past,
* LVEF <50% at screening,
* intolerance to beta-blocker,
* baseline use of any beta-blocker for coronary artery disease including myocardial infarction
* current ACE inhibitor or ARB therapy for hypertension in the presence of diabetes and/or for chronic kidney disease/proteinuria,
* on active therapy with amiodarone, sotalol, or any other antiarrhythmic
* Diagnosis of asthma with current daily use of anti-asthmatic therapy
* heart rate < 50 BPM at screening (average of 3 most recent readings)
* history of or current sick sinus syndrome,
* AV block grade II or higher (unless patient has a permanent pacemaker) at screening,
* systolic blood pressure < 90 mmHg at screening (average of 3 most recent readings)
* severe hepatic dysfunction, as defined by NCI ODWG (total bilirubin >3x ULN, any AST elevation) or Child Pugh C class
* pregnancy
* Metastatic breast cancer (distant metastases)
* Active systemic treatment for non-breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of asymptomatic and symptomatic cardiac dysfunction | 1 year
  Incidence of heart failure or asymptomatic decline in left-ventricular ejection fraction (LVEF) by >10% in patients whose LVEF is ≥50% or LVEF drop ≥5% in those with a decrease to <50% (primary outcome measure)
Rate of reversible cardiac function decline | 1 year
  Reversible LVEF decline to within 5% of baseline (secondary primary outcome measure)

SECONDARY OUTCOMES:
Cardiac function changes after completion of HER2-directed therapy | 1 year
  Delta change in LVEF from completion to one year after completion of trastuzumab-based HER2-directed therapy
Gene variants and risk of cardiotoxicity and response to therapy | 2 years
  Correlation of absolute delta change in GLS and LVEF while on trastuzumab and after stopping trastuzumab with the frequency of the following SNPs: trastuzumab-related: p<1x10-5 hits from Norton GWAS (six loci) 130 HER 2 Ile665Val, HER2 Pro1170Ala125, 126, 130, anthracycline-related: ABCB1 rs1128503, ABCB4 rs1149222, ABCC1 rs45511401, ABCC2 res17222723, CAT rs10836235, CBR3 rs1056892, CYBA rs4673, CYP3A4*22 rs35599367, NCF4 rs1883112, RAC2 rs13058338, RARG rs2229774, SLC28A3 rs7853758, TOP2B rs10865801, and UGT 1A6*4 rs1786378374, 150-152, beta-blocker-related: β2-AR Gln27Gln, β1-AR Arg389Arg 80-82 and CYP2D6 polymorphisms (CYP2D6 alleles (*1, *2, *3, *4, *5, *6, *7, *8, *9, *10, *11, *15, *17, *19, *20, *29, *35, *36, *40 and *41), as well as 7 CYP2D6 gene duplications (*1 9 N, *2 9 N, *4 9 N, *10 9 N, *17 9 N, *35 9 N and *41 9 N) by use of the AmpliChip CYP450 GeneChip

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Herrmann, MD, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials